CLINICAL TRIAL: NCT07315685
Title: Understanding and Treating Severe and Resistant Pathological Aggression: Using Deep Brain Stimulation to Treat Resistant Aggression
Acronym: STAR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Centre Hospitalier du Rouvray (Other Government); Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023/0207/HP; 2025-A00335-44 (Other: IDRCB)
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Autism Spectrum Disorder; Schizophrenia Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Schizophrenia | interventions — Implantable Neurostimulators

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OFF (6-8) ON (8-10) (Experimental): Group 1: stimulation turned off for 2 months (OFF-DBS from M6 to M8) and will be turned back on for 2 months (ON-DBS from M8 to M10).
  Interventions: Device: neurostimulator
- ON (6-8) OFF (8-10) (Experimental): Group 2: stimulation switched on for 2 months (ON-DBS from M6 to M8) and switched off for 2 months (OFF-DBS from M8 to M10).
  Interventions: Device: neurostimulator
- ON (6-7) OFF (7-9) ON (9-10) (Experimental): Group 3: stimulation switched on for 1 month (ON-DBS from M6 to M7), switched off for 2 months (OFF-DBS from M7 to M9) then switched back on for 1 month (ON-DBS from M9 to M10).
  Interventions: Device: neurostimulator

INTERVENTIONS:
Device: neurostimulator — implantation of a neurostimulator and stimulation of the triangle of Sano by alternating ON and OFF phases

SUMMARY:
Physical aggression can be defined as the use of force with the intention of causing physical injury, psychological damage or death. Pathological aggression may be associated with various psychiatric disorders. This symptom can often be improved by prescribing medication, implementing psychoeducational strategies or even electroconvulsive therapy. However, some patients exhibit such severe pathological aggression that they must be institutionalised because they pose a danger to themselves or others. These patients are then hospitalised in a unit for difficult patients (UMD) for enhanced therapeutic care. Despite this maximum level of care, the pathological aggression of a minority of patients persists, leading to a therapeutic impasse, confining the patient to the UMD for many years with social isolation, a collapsed quality of life, and major repercussions for the family. The aim of this project is to use deep brain stimulation, a controlled, reversible, adaptable and low-morbidity neurosurgical method, in six patients with pathological aggression suffering from either schizophrenia (n=3) or autism spectrum disorders (n=3). We hypothesise that the effects of deep brain stimulation (DBS) of the Sano triangle will significantly control the pathological aggression of these six patients.

This is a pilot study with randomised, crossover, double-blind evaluation. It will also provide answers regarding the safety of using SCP for this indication.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 70 inclusive
* Patients who have been in isolation in a secure psychiatric unit for at least 50% of the time over a period of more than 6 months prior to inclusion
* A GAF score <21
* An ICAP score <40
* Other stable medical conditions
* No contraindications to brain imaging (MRI and CT)
* No contraindications to taking medication for travel (loxapine and diazepam)
* No contraindications to surgery
* Adult who has read and understood the information letter and signed the consent form. A psychiatrist, independent of the study and treatment, will examine the patient and determine their ability to read and understand the consent form before signing. If this is not the case, authorisation may be given by the guardianship judge in accordance with Article L. 1111-6.
* An adult assisted by their guardian or by the judge who has read and understood the information letter and signed the consent form (if the patient is under guardianship). If the guardian does not wish to give an opinion or make a decision for the patient, the guardianship judge may be consulted in accordance with Article L1223-1.
* Patients covered by social health insurance (except AME)
* Women of childbearing age (a woman is considered to be of childbearing age, i.e. fertile, after menarche and until she reaches menopause, unless she is permanently infertile) using at least minimally effective contraception (i.e. at least: oral progestogen-only contraception, where inhibition of ovulation is not the primary mode of action, male or female condoms with or without spermicide, diaphragm, diaphragm or sponge with spermicide) for at least 1 month and throughout the study, as well as a negative urinary pregnancy test for β-HCG at inclusion.
* Surgically sterile women (hysterectomy, bilateral salpingectomy and bilateral oophorectomy)
* Menopausal women: Post-menopausal status is defined as the absence of menstruation for 12 months without any other medical cause. Elevated follicle-stimulating hormone (FSH) levels in the post-menopausal interval may be used to confirm post-menopausal status in women who are not using hormonal contraception or hormone replacement therapy. However, in the absence of 12 months of amenorrhoea, a single FSH measurement is insufficient.

For schizophrenic patients

* All previous treatments have failed, including the combination of clozapine (for at least 6 months with clozapine levels > 350 ng/mL) + ECT (minimum 20 sessions)
* Have had at least two clozapine potentiations among the following: lithium, valproic acid, beta-blockers, other antipsychotics.

For ASD patients with or without intellectual disability

- All recommended psychoeducational measures must have been attempted with failure of the following treatments: risperidone, aripiprazole, clozapine, naltrexone, beta-blockers given for at least three months at the maximum tolerated dose.

Exclusion Criteria:

* Minors
* Contraindications to surgery and anaesthesia
* Contraindications to the use of the Medical Device (diathermy, certain magnetic resonance imaging procedures, transcranial magnetic stimulation (TMS), (see section 'Contraindications' in the 'Information for Prescribers' manual for the implanted neurostimulator)
* Contraindications to MRI and CT scans (cardiac or neural pacemakers, ferromagnetic surgical clips, implants and metallic objects, intraocular foreign bodies, pregnancy, claustrophobia, cardiac or neural pacemakers, ferromagnetic surgical clips, implants and metallic objects, intraocular foreign bodies, etc.)
* Other medical problems interfering with the protocol and surgery
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01-13 (Estimated); Primary Completion 2028-10-08 (Estimated); Study Completion 2028-12-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effects of SCP of the Sano triangle on pathological aggression quantified by the MOAS scale after 1 month of SCP compared to the preoperative state. | 9 months

SECONDARY OUTCOMES:
The tolerance and safety of Sano triangle SCP for treating pathological aggression in these six patients, with the collection of potential adverse events, | 10 months
The evaluation of the effects of Sano triangle SCP on pathological behaviours (ICAP scores up to M10), | 10 months
Assessment of the effects of Sano triangle SCP on the number of daily aggressive episodes up to M10 + 1 week, | 10 months
Assessment of the effects of Sano triangle SCP on quality of life (SF-36) up to M10, | 10 months
Assessment of the effects of Sano triangle SCP on socio-familial impact (GAF improved by 20% up to M10), | 10 months
Assessment of the effects of Sano triangle SCP on cognitive and mnemonic impact (TNI-93 up to M10), | 10 months
Study of changes in neuronal activity in local potential fields of the Sano triangle during aggressive episodes up to M10, | 10 months
Anatomical and diffusion MRI study for tractography analysis of fibre bundles in these patients, and study of the volume of activated tissue in relation to the effects observed. | 10 months